CLINICAL TRIAL: NCT02226601
Title: Aprepitant to Mitigate Opioids' Cognitive Side Effects
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Arizona (Other)
Responsible Party: Principal Investigator, Kai Schoenhage, Assistant Professor, University of Arizona
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CognAp
Record Dates: First submitted 2014-08-21; First posted 2014-08-27 (Estimated); Last update posted 2015-06-02 (Estimated); Status verified 2015-05

CONDITIONS: Cognitive Dysfunction
Keywords: drowsiness; loopiness; nausea
MeSH Terms: conditions — Cognitive Dysfunction; Sleepiness; Nausea | interventions — Aprepitant

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Aprepitant (Active Comparator): Aprepitant
  * 40 mg IV pre-operatively
  * 40 mg PO post-op day #1
  * 40 mg PO post-op day #2
  Interventions: Drug: Aprepitant
- Placebo (Placebo Comparator): * electrolyte (0.9% NaCl) infusion) pre-operatively
  * capsule without medication on post-op day #1
  * capsule without medication on post-op day #2
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Aprepitant — 3 days perioperative Aprepitant once a day
  Other Names: Emend
  Arms: Aprepitant
Drug: Placebo — 3 days perioperative Placebot once a day
  Arms: Placebo

SUMMARY:
Morphine and similar substances (called opioids) are often prescribed for moderate to severe pain, such as after a surgery, thus allowing for minimal pain and a better recovery. Unfortunately various, non-dangerous side effects from opioids occur often that limit the way patients feel and can take of themselves, despite otherwise good pain control and minimal limitations from the surgery itself.

DETAILED DESCRIPTION:
In this proposed study the investigators want to examine if the drug aprepitant can decrease the so called "cognitive impairments" opioids may cause, such as drowsiness, loopiness and feeling "high".

This would allow for a better recovery period, in which patients can be more "themselves", participate in activities around them and move forward.

Subjects scheduled for elective surgeries with expected opioid medication for moderate to severe pain and good functional status shortly after surgery will be randomized to receive either aprepitant or placebo shortly before their surgery and for two more days thereafter.

A telephone interview for cognitive status and several specific questions will be used to assess the effect of aprepitant on the subjects' cognitive and functional status.

ELIGIBILITY:
Inclusion Criteria:

* healthy English speaking, opioid-naive consenting adults

Exclusion Criteria:

* current or very recent (< 3 months) opioid therapy
* morbid obesity
* liver disease
* therapy with pimozide, terfenadine, astemizole, cisapride, vitamin K antagonists (warfarin), hormonal contraceptives
* acute or chronic infections
* immunocompromised status
* hemodynamically unstable, hemorrhage (bleeding)
* recent surgery
* pregnancy, nursing
* younger than 18 years old
* not proficient of the English language

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2014-10; Primary Completion 2016-10 (Estimated)

PRIMARY OUTCOMES:
cognitive function | 3 days post-operatively
  questionnaires

CONTACTS AND LOCATIONS:
Overall Officials: Kai Schoenhage, MD, Principal Investigator — University of Arizona
Locations (1):
- University of Arizona Medical Center, Tucson, Arizona, United States

REFERENCES:
- [Background] Walsh SL, Heilig M, Nuzzo PA, Henderson P, Lofwall MR. Effects of the NK1 antagonist, aprepitant, on response to oral and intranasal oxycodone in prescription opioid abusers. Addict Biol. 2013 Mar;18(2):332-43. doi: 10.1111/j.1369-1600.2011.00419.x. Epub 2012 Jan 19. PMID 22260216